CLINICAL TRIAL: NCT02325024
Title: An Open-Label, Single-Dose Study to Compare the Pharmacokinetics (PK) of an Oromucosal Dose of Four Sprays of Sativex® in Subjects With Severe Renal Impairment or End Stage Renal Disease (ESRD), Not Requiring Dialysis, Compared to Matched Subjects With Normal Renal Function.
Brief Title: A Study to Evaluate the Pharmacokinetics Of Sativex® in Subjects With Severe Renal Impairment or End Stage Renal Disease, Compared to Matched Subjects With Normal Renal Function.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: GW Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Organization: GWPharm (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GWCP1426; 2014-003104-67 (EudraCT Number)
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Renal Insufficiency; Kidney Disease
Keywords: Sativex; GW-1000-02; Nabiximols; Pharmacokinetics; Renal Insufficiency; Chronic Kidney Failure
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases; Marijuana Abuse; Kidney Failure, Chronic | interventions — nabiximols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Renally Impaired Subjects (Experimental): Treatment group consists of subjects with severe renal impairment or ESRD and in accordance with the following criteria;
  * Clinically significantly abnormal creatinine and creatinine clearance (CLcr <30 mL/min) and not requiring dialysis.
  * Onset of renal impairment must have been documented at least 3 months prior to study start.
  Interventions: Drug: Sativex
- Matched subjects with Normal Renal Function (Experimental): Group consists of healthy subjects (as determined by medical history, physical examination, biochemistry, hematology, urinalysis, hepatitis B and C, and HIV testing) who demonstrate normal renal function (CLcr > 80 mL/min) and are individually matched to renally impaired subjects with respect to age (within the decile or five years, whichever is less), gender, and Body Mass Index (BMI) (+/- 10% BMI).
  Interventions: Drug: Sativex

INTERVENTIONS:
Drug: Sativex — Each 100 uL actuation (spray) of Sativex contains 27 mg/mL THC and 25 mg/mL CBD plus peppermint flavouring. The study dosage of 10.8 mg THC and 10 mg CBD is delivered as four sprays to the oral mucosa.
  Other Names: GW-1000-02; Nabiximols; THC/CBD spray

SUMMARY:
The study aims to determine the pharmacokinetic (PK) profile of a single oromucosal dose of Sativex® (i.e. how the body absorbs, distributes, metabolises and excretes the drug) when subjects have severe renal impairment or end stage renal disease (ESRD), compared with subjects who have normal renal function.

The primary clinical hypothesis is that there will be an effect from severe renal impairment on the PK of Sativex® when administered as a single oromucosal dose.

The study additionally aims to evaluate the safety and tolerability of the same single oromucosal dose of Sativex® in subjects with severe renal impairment or ESRD.

DETAILED DESCRIPTION:
This is a Phase I, open label, single-dose study to evaluate the effect of renal impairment on the PK of an oromucosal dose (four sprays) of Sativex® (containing 10.8 mg Δ9 tetrahydrocannabinol [THC] and 10 mg cannabidiol [CBD]) in subjects with severe renal impairment or ESRD (with a creatinine clearance < 30 mL/min and not requiring dialysis) compared to matched subjects with normal renal function (with a creatinine clearance > 80 mL/min).

Eligible subjects will be given a single oromucosal dose (four sprays) of Sativex® on Dosing Day 1. Serial blood and urine samples for determination of concentrations of THC, 11-hydroxy- Δ9 - tetrahydrocannabinol (11-OH-THC), CBD, and 7-hydroxy-cannabidiol (7- OH-CBD) will be collected from subjects with severe renal impairment or ESRD, not requiring dialysis, and matched subjects with normal renal function before and up to 48 hours after dosing at selected time points. Pre-dose blood samples will also be collected for protein binding measurement. Safety and tolerability will be evaluated from Day -2 through to the post-study follow-up visit.

The Follow-up Safety visit will be performed 7 days after Sativex® dosing (+ 2 days).

The expected maximum duration for study participation (including Screening, Inpatient Period, and Follow-up) for each individual subject is a maximum of 24 days.

ELIGIBILITY:
Subjects meeting all of the following criteria will be considered eligible for this trial:

General Inclusion Criteria (for all subjects):

1. Willing and able to give written informed consent for participation in the study.
2. Male or female aged 18 years or above.
3. Able (in the investigator's opinion) and willing to comply with all study requirements.
4. Willing and able to communicate with the investigator.
5. Vital signs at screening (after five minutes resting measured in the supine position) within the following ranges:

   1. Body temperature between 35.0-37.5°C
   2. Systolic blood pressure, 90-150 mmHg*
   3. Diastolic blood pressure, 60-90 mmHg*
   4. Pulse rate, 40-99 beats per minute (bpm)*. *Blood pressure and pulse rate will be taken again in a standing position. After two minutes standing, there shall be no more than a 20 mmHg drop in systolic or 10 mmHg drop in diastolic blood pressure, associated with clinical manifestation of postural hypotension.
6. Have a body weight of at least 50.0 kg and have a body mass index (BMI) between 19.0 and 35.0 kg/m2, inclusive.
7. Willing for his or her name to be notified to the responsible authorities for participation in this study, as applicable in individual countries.
8. Willing to allow his or her primary care practitioner and consultant to be notified of participation in the study.

   Inclusion Criteria for Renally Impaired Subjects:
9. Severe renal impairment or ESRD [clinically significantly abnormal creatinine and creatinine clearance (CLcr <30 mL/min and not requiring dialysis].
10. Onset of renal impairment must be documented at least 3 months prior to study start.

    Inclusion Criteria for Normal Renal Function Subjects:
11. In good health as determined by medical history, physical examination, biochemistry, hematology, urinalysis, hepatitis B and C, and HIV testing.
12. Creatinine clearance (CLcr) > 80 mL/min indicating normal renal function.
13. Individually matched to a renally impaired subject with respect to age (within the decile or 5 years, whichever is less), gender, and BMI (+/- 10% BMI).

Exclusion Criteria:

Subjects meeting any of the following criteria will not be eligible for this trial:

1. Donation or loss of 400 mL or more of blood within eight weeks prior to dosing and unwilling to abstain from donation of blood during the study.
2. Significant concomitant illness within the two weeks prior to dosing.
3. At high risk for requiring hospital admission or extended hospital stay during study period or any scheduled elective hospitalization during the planned study duration.
4. Requiring dialysis or expected to require dialysis during study period.
5. Has any surgical or medical condition, significant disease or disorder or any finding on physical examination and/or oral examination (other than their underlying condition) which might significantly alter the absorption, distribution, metabolism or excretion of drugs or that, in the opinion of the investigator, may put the subject at risk, influence the result of the study, or the subject's ability to participate in the study.
6. History of renal transplant.
7. Clinical evidence of acute or chronic liver disease or liver injury as indicated by clinically significant abnormal liver function tests such as Aspartate Aminotransferase, Alanine Aminotransferase, gamma glutamyl-transpeptidase, alkaline phosphatase (any ≥2.5 x Upper Limit of Normal [ULN] ) or serum bilirubin (≥1.5 x ULN) unless there is another likely explanation (e.g. Gilbert's syndrome).
8. Any change in medication within 14 days prior to dosing or planned for anytime throughout the study which might significantly alter the absorption, distribution, metabolism or excretion of the Investigational Medicinal Product (IMP), in the opinion of the investigator.
9. Any known or suspected hypersensitivity to cannabinoids or any of the excipients of the IMP(s).
10. Positive result for the presence of HBsAg, HCAb, or HIV antibodies.
11. Currently using or has used cannabis and/or cannabinoid-based medications (e.g. Marinol®, Nabilone®, Cannador®) within 30 days of study entry and unwilling to abstain for the duration of the study.
12. Any known or suspected history of a substance abuse/dependence disorder within the 12 months prior to dosing or current use of an illicit drug or current non prescribed use of any prescription drug, or evidence of such abuse as indicated by the laboratory assays conducted during the screening or baseline evaluations.
13. Current heavy alcohol consumption (more than 60 g of pure alcohol per day for men, and more than 40 g of pure alcohol per day for women).
14. Unwilling to abstain from drinking alcohol for 24 hours prior to each visit and during the inpatient period of the study.
15. Unwilling to abstain from nicotine products from midnight Day -2 to 48 hours post dose.
16. Unwilling to abstain from grapefruit products for one week prior to and throughout the inpatient period.
17. Consume more than five caffeinated beverages per day (e.g. five cups of tea or coffee or cans of cola) or who are unwilling to abstain from consumption of caffeine-containing food and beverages throughout the inpatient period.
18. Any known or suspected history or immediate family history of schizophrenia, or other psychotic illness, history of severe personality disorder or other severe significant psychiatric disorder other than depression associated with underlying condition.
19. Any history of epilepsy as evidenced by one or more seizures in the last 12 months.
20. Significant cardiac disease, or has a cardiac disorder that in the opinion of the investigator would put the subject at risk of a clinically relevant arrhythmia or myocardial infarction, or has a secondary or tertiary atrioventricular block, or evidence of clinically significant cardiac disease on ECG at screening.
21. Sexually active males whose partner is of childbearing potential who do not agree to practice two different methods of birth control or remain truly abstinent during the study and for three months after the last dose of study medication. Sexually active females of childbearing potential who do not agree to practice two different methods of birth control or remain truly abstinent during the study and for three months after the last dose of study medication. If employing birth control, two of the following precautions must be used: vasectomy, tubal ligation, vaginal diaphragm, intrauterine device, birth control pill, birth control implant, birth control depot injection, condom, or sponge with spermicide. However, a male condom must not be used in conjunction with a female condom as this may not prove effective.

    Note: Non-childbearing potential is defined as female subjects who are surgically sterile (i.e., have undergone bilateral salpingo-oophorectomy, hysterectomy) and female subjects who have been postmenopausal for at least 12 consecutive months.
22. Pregnant, lactating or planning pregnancy during the course of the study and for three months thereafter.
23. Received an IMP within 30 days or five times the half-life of the IMP (whichever is greater) prior to the screening visit.
24. Travel outside the country of residence planned during the study.
25. Previously enrolled into this study or any other Sativex® study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of THC: Cmax, AUC(0-t) and AUC(0-∞) | Pre-dose (t=0) and up to 48 hours post-dose
  The following are presented for THC:
  * Mean maximum (peak) plasma concentration of the drug (Cmax)
  * Mean area under the concentration-time curve calculated to the last observable concentration at time t (AUC(0-t))
  * Mean area under the concentration-time curve from time zero to infinity (AUC(0-∞))
Pharmacokinetic parameters of 11-hydroxy-THC (11-OH-THC): Cmax, AUC(0-t) and AUC(0-∞) | Pre-dose (t=0) and up to 48 hours post-dose
  The following are presented for 11-OH-THC:
  * Mean Cmax
  * Mean AUC(0-t)
  * Mean AUC(0-∞)
Pharmacokinetic parameters of CBD: Cmax, AUC(0-t) and AUC(0-∞) | Pre-dose (t=0) and up to 48 hours post-dose
  The following are presented for CBD:
  * Mean Cmax
  * Mean AUC(0-t)
  * Mean AUC(0-∞)
Pharmacokinetic parameters of 7-hydroxy-CBD (7-OH-CBD): Cmax, AUC(0-t) and AUC(0-∞) | Pre-dose (t=0) and up to 48 hours post-dose
  The following are presented for 7-OH-CBD:
  * Mean Cmax
  * Mean AUC(0-t)
  * Mean AUC(0-∞)

SECONDARY OUTCOMES:
Pharmacokinetic parameters of THC: t(1/2), tmax, CL/F, CLr and F(e,u) | Pre-dose (t=0) and up to 48 hours post-dose
  The following are presented for THC;
  * Mean terminal-phase elimination half-life (t(1/2))
  * Mean time to maximum (peak) plasma concentration (tmax)
  * Mean apparent clearance of drug from plasma (CL/F)
  * Mean renal clearance (CLr)
  * Mean fraction of the systemically available drug excreted into the urine (F(e,u))
Pharmacokinetic parameters of 11-OH-THC: t(1/2), tmax, CLr and F(e,u) | Pre-dose (t=0) and up to 48 hours post-dose
  The following are presented for 11-OH-THC;
  * Mean t(1/2)
  * Mean tmax
  * Mean CLr
  * Mean F(e,u)
Pharmacokinetic parameters of CBD: t(1/2), tmax, CL/F, CLr and F(e,u) | Pre-dose (t=0) and up to 48 hours post-dose
  The following are presented for CBD;
  * Mean t(1/2)
  * Mean tmax
  * Mean CL/F
  * Mean CLr
  * Mean F(e,u)
Pharmacokinetic parameters of 7-OH-CBD: t(1/2), tmax, CLr and F(e,u) | Pre-dose (t=0) and up to 48 hours post-dose
  The following are presented for 7-OH-CBD;
  * Mean t(1/2)
  * Mean tmax
  * Mean CLr
  * Mean F(e,u)
Pharmacokinetic parameters of THC: Cmax(u), AUC(0-t(u)), AUC(0-∞(u)) and CLu/F | Pre-dose (t=0) and up to 48 hours post-dose
  The following are presented for THC:
  * Mean unbound maximum (peak) plasma concentration of the drug (Cmax(u))
  * Mean unbound area under the concentration-time curve calculated to the last observable concentration at time t (AUC(0-t(u)))
  * Mean unbound area under the concentration-time curve from time zero to infinity (AUC(0-∞(u)))
  * Mean apparent unbound clearance of drug from plasma (CLu/F)
Pharmacokinetic parameters of 11-OH-THC: Cmax(u), AUC(0-t(u)) and AUC(0-∞(u)) | Pre-dose (t=0) and up to 48 hours post-dose
  The following are presented for 11-OH-THC:
  * Mean Cmax(u)
  * Mean AUC(0-t(u))
  * Mean AUC(0-∞(u))
Pharmacokinetic parameters of CBD: Cmax(u), AUC(0-t(u)), AUC(0-∞(u)) and CLuF | Pre-dose (t=0) and up to 48 hours post-dose
  The following are presented for CBD:
  * Mean Cmax(u)
  * Mean AUC(0-t(u))
  * Mean AUC(0-∞(u))
  * Mean CLu/F
Pharmacokinetic parameters of 7-OH-CBD: Cmax(u), AUC(0-t(u)) and AUC(0-∞(u)) | Pre-dose (t=0) and up to 48 hours post-dose
  The following are presented for 11-OH-THC:
  * Mean Cmax(u)
  * Mean AUC(0-t(u))
  * Mean AUC(0-∞(u))
The incidence of adverse events as a measure of subject safety | From screening to follow-up (a maximum of 24 days)
  The number of subjects who experienced an adverse event during the study is presented. The time-frame for adverse event reporting was from screening to the follow-up visit.
The number of subjects with a clinically significant change in physical and oral examination results, relative to pre-treatment baseline | From screening to follow-up (a maximum of 24 days)
  The number of subjects with a change in physical and oral examination results indicative of an adverse event, relative to the pre-treatment baseline, is presented.
The number of subjects with a clinically significant change in 12-lead electrocardiogram (ECG) results, relative to pre-treatment baseline | From screening to follow-up (a maximum of 24 days)
  The number of subjects with a change in ECG results indicative of an adverse event, relative to the pre-treatment baseline, is presented.
The number of subjects with clinically significant changes in laboratory test parameters, relative to pre-treatment baseline | From screening to follow-up (a maximum of 24 days)
  The number of subjects with clinically significant changes in serum biochemistry, hematology and urinalysis, relative to the pretreatment baseline, is presented.
The number of subjects with a clinically significant change in vital signs, relative to pre-treatment baseline | From screening to follow-up (a maximum of 24 days)
  The number of subjects with a clinically significant change in vital signs (systolic blood pressure, diastolic blood pressure, pulse rate) indicative of an adverse event, relative to the pre-treatment baseline, is presented.
  A clinically significant drop in blood pressure is defined as a 20 mmHg drop in systolic or 10 mmHg drop in diastolic blood pressure associated with a clinical manifestation of postural hypotension after two minutes standing.